CLINICAL TRIAL: NCT02588144
Title: Combined Stimulation of Subthalamic Nucleus and Substantia Nigra Pars Reticulata for Resistant Freezing of Gait in Parkinson's Disease: A Randomized Controlled Multicenter Trial
Brief Title: Combined Stimulation of STN and SNr for Resistant Freezing of Gait in Parkinson's Disease
Acronym: STN+SNr
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Daniel Weiss, MD, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IHanci
Record Dates: First submitted 2015-10-24; First posted 2015-10-27 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; freezing of gait; deep brain stimulation; substantia nigra pars reticulata; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- [standard STN] (Active Comparator): Device: standard stimulation on subthalamic (STN) contacts
  Interventions: Procedure: [standard STN]
- [STN+SNr] (Experimental): Device: Combined stimulation of the subthalamic nucleus (STN) and the substantia nigra pars reticulata (SNr)
  Interventions: Procedure: [STN+SNr]

INTERVENTIONS:
Procedure: [standard STN] — High frequency deep brain stimulation with variable (best individual) stimulation on subthalamic contacts
  Other Names: subthalamic deep brain stimulation
  Arms: [standard STN]
Procedure: [STN+SNr] — high frequency deep brain stimulation of combined (best individual) subthalamic and nigral stimulation
  Other Names: combined subthalamic and nigral stimulation
  Arms: [STN+SNr]

SUMMARY:
54 patients with idiopathic Parkinson's disease and freezing of gait resistant to subthalamic nucleus stimulation and dopaminergic medication will be included into this multicentre randomised controlled double-blinded parallel group clinical trial. The treatment consists of two different stimulation settings using (i) conventional stimulation of the subthalamic nucleus [standard STN] as active comparator and (ii) combined stimulation of active electrode contacts located in both the subthalamic nucleus and substantia nigra pars reticulata [STN+SNr].

DETAILED DESCRIPTION:
The primary endpoint of this study is to investigate the efficacy and safety of combined [STN+SNr] stimulation by "interleaving stimulation" as compared to [standardSTN] after 3 months on refractory freezing of gait (FOG). The Trial is designed as superiority study with an 80% power to detect a mean improvement of 4.7 points on the Freezing of Gait Assessment Course (Ziegler et al., 2010) with one-tailed P < 0.2. To this end 54 patients will be studied. After a common baseline assessment in [standardSTN], patients will be randomized to either [standardSTN] or [STN+SNr] in 1:1 ratio (27 per arm). The primary endpoint assessment is scheduled 90 days from baseline assessment (V6). Additional interim visits are scheduled for secondary purpose from baseline at day 2 (V2), day 8 (V3), day 21 (V4), day 42 (V5).

The rationale for this study comes from our previous phase II trial (Weiss et al., 2013) in which we have observed an improvement of freezing of gait from combined STN+SNr stimulation as secondary endpoint compared with standard STN stimulation at three-week follow-up.

Secondary outcome measures include anamnestic assessments on freezing of gait and falls, balance, quality of life, neuropsychiatric symptoms and suicidality.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (according to the "British Brain Bank criteria" (Hughes, 1992) including genetic forms
* Therapy with STN-DBS (deep brain stimulation) (ACTIVA pulse generators) at least six months from surgery
* Activa PC (Primary Cell) or Activa RC (Rechargeable Cell) as implanted pulse generator with "Interleaving" programming option
* Localization of an active electrode contact in the subthalamic nucleus
* Localization of the caudal electrode contacts in the substantia nigra pars reticulata area (coordinates relative to midcommisural Point (MCP):

left: -7mm ≤ x ≤ -12mm; -2mm ≤ y ≤ -6mm; -6mm ≤ z ≤ -10mm right: 7mm ≤ x ≤ 12mm; -2mm ≤ y ≤ -6mm; -6mm ≤ z ≤ -10mm (x = medio-lateral, y = anterio-posterior, z = rostro-caudal)

* ≥ 30% improvement in UPDRS III with 'standard STN' compared to 'stimulation off' in dopaminergic off
* Freezing of Gait Assessment Course ≥10 and ≤33
* Patient not wheelchair-bound and possible to move self-dependently outside a freezing episode.
* Disease duration ≥ 5 years
* Age: between 18 and 80 years
* Dopaminergic medication constant for at least four weeks prior to study enrolment
* Written informed consent

Exclusion Criteria:

* Participation in other clinical trials within the past three months and during enrolment in our study
* Cognitive impairment (Mini Mental State Exam < 20)
* Suicidality, Psychosis
* Other severe pathological chronic condition that might confound treatment effects or interpretation of the data
* Pregnancy
* Paradoxical levodopa-induced "on" state freezing (Espay et al., 2012)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Freezing of Gait Assessment Course (FOG-AC) | Outcome at day 90 (V6) with reference to baseline (V1)

SECONDARY OUTCOMES:
Timed Walking test from Core Assessment Program for Surgical Interventions in Parkinson's disease (CAPSIT-PD) | At baseline, day 2, 8, 21, 42 and 90, respectively
Berg Balance Scale | At baseline, day 42 and 90, respectively
Parkinson's disease questionnaire (PDQ-39) | At baseline, day 42 and 90, respectively
Freezing of gait questionnaire | At baseline, day 42 and 90, respectively
Beck's depression Inventory | At baseline, day 42 and 90, respectively
Columbia-Suicide Severity Rating Scale | At baseline, day 42 and 90, respectively
Clinical global impression scale | At day 42 and 90, respectively
Falls diary | At baseline, day 2, 8, 21, 42 and 90, respectively
Movement Disorders Society Unified Parkinson's disease Rating Scale (MDS-UPDRS III) | At baseline, day 2, 8, 21, 42 and 90, respectively
Movement Disorders Society Unified Parkinson's disease Rating Scale (MDS-UPDRS II) | At baseline, day 42 and 90, respectively
Movement Disorders Society Unified Parkinson's disease Rating Scale (MDS-UPDRS IV) | At baseline, day 42 and 90, respectively
Freezing of Gait Assessment Course (FOG-AC) | At baseline, day 2, 8, 21, 42 after active treatment (STN vs. STN+SNr), respectively
  To determine treatment kinematics

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, MD, Principal Investigator — Department for Neurodegenerative Diseases, Centre for Neurology, Tübingen, Germany, and Hertie-Institute for Clinical Brain Research; Alireza Gharabaghi, MD, Principal Investigator — Division of Functional and Restorative Neurosurgery, Department of Neurosurgery, Tübingen, Germany, and Center for Integrative Neuroscience, Tübingen, Germany
Locations (10):
- Germany (9):
  - Center of Neurology and Hertie Institute for Clinical Brain Research, Department for Neurodegenerative Diseases and Neurosurgery University of Tübingen, Tübingen, Baden-Wurttemberg
  - Ludwig-Maximilians-University Munich, Klinikum Großhadern, Department for Neurology and Neurosurgery, Munich, Bavaria
  - University Hospital Regensburg , Department for Neurology and Neurosurgery, Regensburg, Bavaria
  - University Hospital Köln, Department for Neurology and Neurosurgery, Cologne, North Rhine-Westphalia
  - University Hospital of Düsseldorf, Departments for Neurology and Neurosurgery, Düsseldorf, North Rhine-Westphalia
  - University Hospital Leipzig, Department for Neurology and Neurosurgery, Leipzig, Saxony
  - University Hospital Kiel, Department for Neurology and Neurosurgery, Kiel, Schleswig-Holstein
  - Charite- University Hospital Berlin, Departments for Neurology and Neurosurgery, Berlin
  - University Hospital Hamburg-Eppendorf, Department for Neurology and Neurosurgery, Hamburg
- University Hospital Luxembourg, Department for Neurology and Neurosurgery, Luxembourg, Luxembourg

REFERENCES:
- [Result] Weiss D, Walach M, Meisner C, Fritz M, Scholten M, Breit S, Plewnia C, Bender B, Gharabaghi A, Wachter T, Kruger R. Nigral stimulation for resistant axial motor impairment in Parkinson's disease? A randomized controlled trial. Brain. 2013 Jul;136(Pt 7):2098-108. doi: 10.1093/brain/awt122. Epub 2013 Jun 11. PMID 23757762